CLINICAL TRIAL: NCT03462563
Title: A Prospective, Multicenter, Randomized Controlled Study to Evaluate the Effect of GYNECARE INTERCEED™ Absorbable Adhesion Barrier in Preventing the Abdominal Incision Adhesions
Brief Title: Prospective, Multicenter, Randomized Controlled Study to Evaluate the Effect of INTERCEED™
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because the pre-specified study stopping criterion has been met.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESC-201701
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Subjects Scheduled to Undergo Laparoscopic Radical Resection of Rectal Carcinoma With Preventive Ileostomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERCEED™ (Experimental): patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo). In subjects assigned to the treatment arm, the INTERCEED™ must be applied beneath the target incision site (the midline incision mainly for the removal specimen).
  Interventions: Device: INTERCEED™
- standard of care treatment (Placebo Comparator): During the Phase 1 operation, when the definite decision to create a temporary ostomy is made, patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo).
  Interventions: Device: Placebo

INTERVENTIONS:
Device: INTERCEED™ — when the definite decision to create a temporary ostomy is made, patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo). In subjects assigned to the treatment arm, the INTERCEED™ must be applied beneath the target incision site (the midline incision mainly for the removal specimen)
  Arms: INTERCEED™
Device: Placebo — During the Phase 1 operation, when the definite decision to create a temporary ostomy is made, patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo).
  Arms: standard of care treatment

SUMMARY:
This is a prospective, randomized controlled study. The study population will include 220 subjects scheduled to undergo laparoscopic radical resection of rectal carcinoma with preventive ileostomy (Phase 1 operation).

During the Phase 1 operation, when the definite decision to create a temporary ostomy is made, patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo). In subjects assigned to the treatment arm, the INTERCEED™ must be applied beneath the target incision site (the midline incision mainly for the removal specimen). The subjects will return 3-9 months after the phase 1 operation (colorectal resection with temporary ileostomy) for phase 2 operation, to have their diverting ostomy taken down (ileostomy reversal). During the phase 2 operation (ileostomy reversal), the incidence, extent and severity of adhesions will be evaluated through the laparoscope.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study. The study population will include 220 subjects scheduled to undergo laparoscopic radical resection of rectal carcinoma with preventive ileostomy (Phase 1 operation).

During the Phase 1 operation, when the definite decision to create a temporary ostomy is made, patients will be randomized in 1:1 ratio to either the treatment arm (INTERCEED™) or the control arm (standard of care treatment: no adhesion barrier, no placebo). In subjects assigned to the treatment arm, the INTERCEED™ must be applied beneath the target incision site (the midline incision mainly for the removal specimen).

The subjects will return 3-9 months after the phase 1 operation (colorectal resection with temporary ileostomy) for phase 2 operation, to have their diverting ostomy taken down (ileostomy reversal).

During the phase 2 operation (ileostomy reversal), the incidence, extent and severity of adhesions will be evaluated through the laparoscope.

An ad-hoc interim analysis is proposed based on feedback received from the investigators who observed very low rate of adhesions at the second procedure for ostomy reversal. The ad-hoc interim analysis is planned to be performed while at least 61% of the total number of participants with evaluable primary endpoints are available. If the conditional power (CP) is ≤ 60%, the observed adhesion rate difference magnitude is much less than the assumed difference magnitude of 0.25, therefore, the study will be terminated due to low adhesion rate and small effect size between INTERCEED and control arms. Otherwise, the study will continue until the study completion as planned.

ELIGIBILITY:
Inclusion Criteria:

Subjects elder than 18 years of age who require laparoscopic colorectal resection with the formation of a temporary diverting loop ileostomy and a planned closure of diverting ileostomy within 3 to 7 months The subjects should be willing to participate in the study, comply with study requirements, follow-up schedule, and give written informed consent prior to any study-related procedures The target incision length less than 8cm allowing the INTERCEED (product length 10.2cm) to overlap at least 1cm beyond each pole of the incision The subject is believed to have life expectancy more than 12 months after Phase 1 operation, based on investigators assessment.

Exclusion Criteria Female patients who are pregnant or lactating at the time of screening Patient with a history of mechanical bowel obstruction but except the mechanical bowel obstruction caused by the colorectal cancer treated in the Phase I operation. Subjects with history of mid and lower abdominal region or pelvic surgery Patients for whom it is known that loop ileostomy closure within 3 to 9 months is not feasible Patients with a history of active intra-abdominal infection such as peritonitis or abdominal abscess Patients with a history of intestinal fistulae Patients with a history of endometriosis Intended use of intraoperative lavage/irrigation with any anti-adhesion solutions other than saline or an adhesion barrier other than INTERCEED Use of immune system suppressants deemed by the investigator to interfere with wound healing Impaired immune system function or coagulation disorders deemed by the surgeon to interfere with wound healing.

Bevacizumab use within 30 days prior to surgery Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedures Patients with evidence of distant metastasis of the primary colorectal cancer Patients who underwent abdominal radiotherapy before Phase 1 operation Adhesions (Grade 2-3 adhesion) and/or gross contamination (caused by tumor perforation) present in the abdominal cavity at the Phase 1 operation The rectal carcinoma radical resection (R0 resection) preventive ileostomy are not performed in Phase 1 operation pected resection of other organs (bladder, uterus) during Phase 1 operation Use of topical haemostatic products, local motherapeutic products or other drugs and/or medical device in abdominal/pelvic cavity which may impact the study primary endpoint judged by the investigator Patient is participating in other investigational drug or device study within 30 days or 5 half-lives of an investigational drug A known history of severe multiple drug allergies or known allergy to cellulose or cellulose derived products Any medications, treatments and/or implanted devices (except INTERCEED) that on investigator's opinion may be adhesiogenic or may potentially affect the observation of postoperative adhesions Any physical or psychological conditions that at discretion of investigators may impair study participation A medical condition or other serious conditions that will interfere with compliance and/or ability to complete this study protocol; or Any other situation or reason that at discretion of investigators is unsuitable for study participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - First affiliated hospital of zhengzhou university, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The 2nd affiliated Hospital of Zhongnan University, Changsha, Hunan
  - The affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shanghai Jiaotong University School of Medcine, Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Chinese PLA General Hospital, Beijing
  - Friendship Hospital, Beijing
  - Changhai Hospital, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: INTERCEED: In participants assigned to the treatment arm, the INTERCEED was applied beneath the target incision site (the midline incision for the removal specimen) (Phase 1 operation). After 3-9 months of Phase 1 operation, participants undergo ileostomy reversal (Phase 2 operation).
- Control Arm: Standard of Care (SOC): Participants received standard of care treatment: no adhesion barrier, no placebo (Phase 1 operation).
Period: Overall Study
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Started | 94 | 81
Completed | 79 | 64
Not Completed | 15 | 17
Not completed — Death | 1 | 1
Not completed — Termination of study | 2 | 1
Not completed — Adverse Event | 1 | 3
Not completed — Unspecified reason | 10 | 12
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) set contained all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC) | Total
Number analyzed (Participants) | 94 | 81 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.30) | 59.7 (9.34) | 58.2 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 72 | 57 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 93 | 78 | 171
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 94 | 81 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free of Adhesions at the Target Incision Site
Description: Percentage of participants free of adhesions at the target incision site in each study group based on evaluation through laparoscopy at ileostomy reversal were reported.
Time Frame: 3 to 9 months after phase 1 operation
Population: The Intent-to-treat (ITT) set contained all randomized participants. Here "N" (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 72 | 60
percentage of participants | 86.1 | 86.7

2. Secondary Outcome: Number of Participants With Extent of Adhesions at Target Incision Site in Phase 2 Operation
Description: Number of participants with extent of adhesions at target incision site in Phase 2 operation were reported. The extent of adhesions (percentage of the area covered by adhesion) was evaluated based on Grade 1: mild, covering up to 25 percent (%) of the total area and length; Grade 2: moderate, covering 26%-50% of the total area and length; and Grade 3: severe, covering over 50% of the total area and length.
Time Frame: 3 to 6 months after phase 1 operation
Population: The ITT set contained all randomized participants. Here "N" (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 72 | 60
Participants
  No adhesion | 62 | 52
  Grade 1 | 5 | 3
  Grade 2 | 3 | 1
  Grade 3 | 2 | 4

3. Secondary Outcome: Number of Participants With Severity of Adhesions at Target Incision Site in Phase 2 Operation
Description: Number of participants with severity of adhesions at target incision site in Phase 2 operation were reported. The severity of adhesions was evaluated based on Grade 1: filmy thickness, avascular; Grade 2: moderate thickness, limited vascularity and Grade 3: dense thickness, vascularized.
Time Frame: 3 to 9 months after phase 1 operation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 72 | 59
Participants
  No adhesion | 62 | 52
  Grade 1 | 7 | 2
  Grade 2 | 3 | 5
  Grade 3 | 0 | 0

4. Secondary Outcome: Number of Participants With Extent of Adhesions at Four Abdominal Quadrants in Phase 2 Operation
Description: Number of participants with extent of adhesions at four abdominal quadrants in Phase 2 operation were reported. The abdominal cavity was divided into four abdominal quadrants as: Right upper abdominal quadrant, Left upper abdominal quadrant, Right lower abdominal quadrant and Left lower abdominal quadrant and the extent of adhesions (percentage of the area covered by adhesion) was evaluated based on Grade 1: mild, covering up to 25% of the total area and length; Grade 2: moderate, covering 26%-50% of the total area and length; and Grade 3: severe, covering over 50% of the total area and length. One participant may have multiple sites of adhesion.
Time Frame: 3 to 9 months after phase 1 operation
Population: The ITT set contained all randomized participants. Here "N" (number of participants analyzed) signifies participants who were evaluated for this outcome measure. Here "n" (number analyzed) signifies participants who were evaluated for a specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 25 | 29
Participants
  Right Upper Abdominal Quadrant: Grade 1: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 1 | 7 | 9
  Right Upper Abdominal Quadrant: Grade 2: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 2 | 1 | 0
  Right Upper Abdominal Quadrant: Grade 3: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 3 | 0 | 0
  Left Upper Abdominal Quadrant: Grade 1: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 1 | 3 | 6
  Left Upper Abdominal Quadrant: Grade 2: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 2 | 1 | 0
  Left Upper Abdominal Quadrant: Grade 3: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 3 | 0 | 0
  Right Lower Abdominal Quadrant: Grade 1: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 1 | 11 | 12
  Right Lower Abdominal Quadrant: Grade 2: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 2 | 1 | 1
  Right Lower Abdominal Quadrant: Grade 3: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 3 | 0 | 0
  Left Lower Abdominal Quadrant: Grade 1: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 1 | 10 | 10
  Left Lower Abdominal Quadrant: Grade 2: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 2 | 0 | 0
  Left Lower Abdominal Quadrant: Grade 3: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 3 | 0 | 0

5. Secondary Outcome: Number of Participants With Severity of Adhesions at Four Abdominal Quadrants in Phase 2 Operation
Description: Number of participants with severity of adhesions at four abdominal quadrants in Phase 2 operation were reported. The abdominal cavity was divided into four abdominal quadrants as: Right upper abdominal quadrant, Left upper abdominal quadrant, Right lower abdominal quadrant and Left lower abdominal quadrant and the severity of adhesions was evaluated based on Grade 1: filmy thickness, avascular; Grade 2: moderate thickness, limited vascularity and Grade 3: dense thickness, vascularized. One participant may have multiple sites of adhesion.
Time Frame: 3 to 6 months after phase 1 operation
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 25 | 29
Participants
  Right Upper Abdominal Quadrant: Grade 1: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 1 | 7 | 8
  Right Upper Abdominal Quadrant: Grade 2: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 2 | 1 | 1
  Right Upper Abdominal Quadrant: Grade 3: number analyzed (Participants) | 8 | 9
  Right Upper Abdominal Quadrant: Grade 3 | 0 | 0
  Left Upper Abdominal Quadrant: Grade 1: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 1 | 3 | 6
  Left Upper Abdominal Quadrant: Grade 2: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 2 | 1 | 0
  Left Upper Abdominal Quadrant: Grade 3: number analyzed (Participants) | 4 | 6
  Left Upper Abdominal Quadrant: Grade 3 | 0 | 0
  Right Lower Abdominal Quadrant: Grade 1: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 1 | 11 | 10
  Right Lower Abdominal Quadrant: Grade 2: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 2 | 1 | 3
  Right Lower Abdominal Quadrant: Grade 3: number analyzed (Participants) | 12 | 13
  Right Lower Abdominal Quadrant: Grade 3 | 0 | 0
  Left Lower Abdominal Quadrant: Grade 1: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 1 | 10 | 10
  Left Lower Abdominal Quadrant: Grade 2: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 2 | 0 | 0
  Left Lower Abdominal Quadrant: Grade 3: number analyzed (Participants) | 10 | 10
  Left Lower Abdominal Quadrant: Grade 3 | 0 | 0

6. Secondary Outcome: Number of Participants With Mechanical Ileus
Description: Number of participants with mechanical ileus were reported. Incidence of mechanical ileus was defined as the mechanical ileus judged by investigators, which occurred 1 week after Phase 1 operation. Incidence of mechanical ileus was reported based on three categories: Post-Phase 1 operation through 7 days after Phase 1 operation (less than or equal to [<=] 7 days) (for participants underwent Phase 1 operation), 7 days after Phase 1 operation through pre-Phase 2 operation (for participants underwent Phase 1 operation) and Post-Phase 2 operation (for participants underwent Phase 2 operation).
Time Frame: Up to 9 months after phase 1 operation
Population: The Safety Set (SS) contained all participants who were treated with study product or control (no adhesion barrier) as per the protocol. Here "n" (number analyzed) is defined as the number of participants evaluable for a specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
Number analyzed (Participants) | 93 | 81
Participants
  Post-Phase 1 Operation Through 7 Days After Phase 1 Operation (<=7 days) | 3 | 1
  7 Days After Phase 1 Operation Through pre-Phase 2 Operation | 1 | 0
  Post-Phase 2 Operation (for Participants Underwent Phase 2 Operation): number analyzed (Participants) | 79 | 65
  Post-Phase 2 Operation (for Participants Underwent Phase 2 Operation) | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 9.5 months
Description: The Safety Set (SS) contained all participants who were treated with study product or control (no adhesion barrier) as per the protocol.
Arm/Group | Treatment Arm: INTERCEED | Control Arm: Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 1/93 | 1/81
Serious Adverse Events (participants affected / at risk) | 21/93 | 26/81
Other Adverse Events (participants affected / at risk) | 61/93 | 44/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm: INTERCEED (N=93) | Control Arm: Standard of Care (SOC) (N=81)
Anastomotic leak (Injury, poisoning and procedural complications) | 2 | 2
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Stoma site oedema (Injury, poisoning and procedural complications) | 1 | 0
Stoma site dermatitis (Injury, poisoning and procedural complications) | 0 | 1
Stoma obstruction (Injury, poisoning and procedural complications) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Subileus (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pelvic infection (Infections and infestations) | 1 | 2
Postoperative wound infection (Infections and infestations) | 1 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Aortic disorder (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Decreased immune responsiveness (Immune system disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm: INTERCEED (N=93) | Control Arm: Standard of Care (SOC) (N=81)
Stomal hernia (Injury, poisoning and procedural complications) | 12 | 11
Incision site pain (Injury, poisoning and procedural complications) | 12 | 7
Wound complication (Injury, poisoning and procedural complications) | 3 | 5
Stoma complication (Injury, poisoning and procedural complications) | 2 | 3
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hypertension (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1
Vomiting (Gastrointestinal disorders) | 12 | 5
Nausea (Gastrointestinal disorders) | 9 | 3
Abdominal distension (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Retching (Gastrointestinal disorders) | 2 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 21 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Acute phase reaction (General disorders) | 16 | 8
Localised oedema (General disorders) | 1 | 2
Pain (General disorders) | 1 | 2
Hyperthermia (General disorders) | 0 | 2
Chills (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Urine output decreased (Investigations) | 5 | 3
Blood albumin decreased (Investigations) | 4 | 4
Blood pressure increased (Investigations) | 3 | 4
Platelet count decreased (Investigations) | 3 | 3
C-reactive protein increased (Investigations) | 2 | 3
Neutrophil count increased (Investigations) | 2 | 3
Weight decreased (Investigations) | 0 | 5
White blood cell count decreased (Investigations) | 2 | 3
White blood cell count increased (Investigations) | 1 | 2
Heart rate increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 1 | 1
Neutrophil percentage increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Red blood cells urine positive (Investigations) | 1 | 0
Cardiac function test abnormal (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0
Carbohydrate antigen 125 increased (Investigations) | 1 | 0
Granulocyte count decreased (Investigations) | 1 | 0
Tumour marker increased (Investigations) | 1 | 0
Lipids increased (Investigations) | 1 | 0
Nutritional condition abnormal (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Blood test abnormal (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Procalcitonin abnormal (Investigations) | 0 | 1
Bone scan abnormal (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 8
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Small airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 6 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 2
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 5 | 6
Oliguria (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Bladder irritation (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hypotension (Vascular disorders) | 3 | 3
Hypertension (Vascular disorders) | 3 | 3
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 1
Listless (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Hyperplasia adrenal (Endocrine disorders) | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 1
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 2
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Stoma site oedema (Injury, poisoning and procedural complications) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Myelosuppression (Blood and lymphatic system disorders) | 4 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pelvic infection (Infections and infestations) | 1 | 2
Postoperative wound infection (Infections and infestations) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 11

LIMITATIONS AND CAVEATS:
The study was terminated due to small effect size between INTERCEED and control arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT03462563/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03462563/SAP_001.pdf